CLINICAL TRIAL: NCT04514510
Title: A Study to Evaluate the Effects of Fixed Dose Flavonoid Isoquercetin on Thrombo-Inflammatory Biomarkers in Subjects With Stable Sickle Cell Disease
Brief Title: Fixed Dose Flavonoid Isoquercetin on Thrombo-Inflammatory Biomarkers in Subjects With Stable Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Quercis Pharma AG (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200137; 20-H-0137
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-11

CONDITIONS: Sickle Cell Disease
Keywords: Venous thrombosis; Protein disulfide isomerase; Thrombo-inflammation; HbS polymerization; P-selectin
MeSH Terms: conditions — Anemia, Sickle Cell; Venous Thrombosis | interventions — isoquercitrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with Sickle Cell Disease Receiving Isoquercetin (Experimental): Isoquercetin 1000 mg, once daily by mouth for 28 days in participants with Sickle Cell Disease.
  Interventions: Drug: Isoquercetin
- Participants with Sickle Cell Disease Receiving Placebo (Placebo Comparator): Placebo once daily, by mouth for 28 days in participants with Sickle Cell Disease.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isoquercetin — Isoquercetin (quercetin-3-O-beta-D-glucoside, also referred to as isoquercitrin) is a naturally occurring monoglucoside of the most studied and widely consumed bioflavonoid, quercetin.
  Isoquercetin given at 1000 mg, once daily by mouth for 28 days.
  Other Names: isoquercitrin
  Arms: Participants with Sickle Cell Disease Receiving Isoquercetin
Drug: Placebo — Silicified microcrystalline cellulose NF, Ascorbic acid, Nicotinic acid, Mg stearate, Silica and Colloidal Anhydrous Ph. Eur./Colloidal Silicon dioxide USP/NF.
  Placebo give at 1000 mg, once daily by mouth for 28 days.
  Arms: Participants with Sickle Cell Disease Receiving Placebo

SUMMARY:
Background:

Sickle cell disease (SCD) is an inherited hemoglobin disorder. People with SCD have an increased chance for getting blood clots. Researchers want to see if a dietary supplement called isoquercetin can decrease levels of inflammation and blood clotting in people with SCD.

Objective:

To see how isoquercetin works in people with SCD.

Eligibility:

Adults age 18-70 years old who have SCD and are in a steady-state (have not experienced a pain crisis in the last 60 days and, if taking hydroxyurea, have not had a dose change in the past 90 days).

Design:

Participants will be screened with a physical exam, medical history, medicine review, and blood tests.

Participants will be put in 1 of 2 treatment groups. They will take 4 capsules of isoquercetin or placebo all at once, by mouth, every day for 4 weeks. They will get a pill dispenser and keep a medicine diary.

Participants may have an optional near infrared spectroscopy (NIRS) test to measure how treatment affects blood flow. In this test, probes will be placed on the skin to measure tissue oxygen level and blood flow. A blood pressure cuff placed on the arm will be filled with air briefly to restrict the blood flow in the arm (for up to 5 minutes) and then released. Participants may also be asked to breathe at a certain rate or hold their breath for as long as they can during measurements.

Participants will take folic acid once a day.

Participants will have an end-of-study drug visit. They will discuss any side effects and repeat some of the screening tests. They may have an additional optional NIRS test.

About a month after the end of study drug visit, participants will be contacted by phone to see if they have any side effects. Those who do may have a follow-up visit. At this visit, they may have additional blood tests performed.

Participation will last from 8 to 12 weeks.

DETAILED DESCRIPTION:
Sickle Cell Disease (SCD) is an inherited monogenic hemoglobin disorder caused by a mutation in the gene encoding the beta globin subunit of adult hemoglobin (HbA) resulting in a substitution of valine for glutamic acid at position 6 and thus producing hemoglobin S (HbS). When deoxygenated, HbS polymerizes, rendering the red cell rigid, viscous, and abnormally adherent to the capillary endothelium. This impedes blood flow in the microcirculation, causing ischemia and microinfarcts that lead to painful crises, cerebrovascular stroke, renal impairment, venous blood clots, retinopathy and other end-organ damage. The current scientific literature recognizes the contribution of an acquired hypercoagulable state in SCD to vascular pathobiology, chronic organ dysfunction, and mortality.

Like cancer, SCD is associated with a hypercoagulable state and patients have a high risk of new onset and recurrent venous thromboembolism (VTE). Elevated blood levels of the procoagulant protein tissue factor and its activator, protein disulfide isomerase (PDI) in patients with SCD suggest a causal role for these proteins in the development of venous blood clots. In cancer patients, inhibiting plasma PDI activity with isoquercetin (IQ) led to a significant reduction in VTE biomarkers (soluble P-selectin and D-dimer) and venous thrombosis over the short term. These findings provide support to test the hypothesis that isoquercetin treatment in sickle cell disease would diminish thrombo-inflammatory biomarkers and attenuate the hypercoagulable state.

ELIGIBILITY:
* INCLUSION CRITERIA:

For enrollment onto the active phase of the study (IQ supplement vs placebo), subjects must meet all of the following criteria during the screening period (visit #1) which can last from 0-28 days prior to start of study intervention:

* Unequivocal diagnosis of sickle cell anemia (Hemoglobin SS or Hemoglobin SC or Beta Thalassemia Major or Beta Thalassemia Minor) confirmed by hemoglobin electrophoresis performed on patients at least 90 days after a blood transfusion if previously transfused, or DNA genotyping.
* Age 18-70 years old
* Steady state SCD (no acute vaso-occlusive crisis within 60 days of D0 of the study) and if on HU therapy, on an optimized dose for at least 30 days. For those newly initiated on HU therapy, the dose should be unchanged for at least 90 days.
* Be willing to comply with all study procedures for the duration of the study.
* Have provided signed written informed consent prior to performing any study procedure, including screening procedures.

EXCLUSION CRITERIA:

Subjects who meet any of the following criteria during screening will not receive the study intervention and will be counted toward study accrual. Screen failures will not be included in the analysis for statistical purposes:

* SCD with a recent VOC (<60 days from D0 of study).
* SCD with history of recent blood transfusion (<60 days from D0 of study) or exchange transfusion (<90 days from D0 of study).
* SCD with a recent VTE (within 90 days of diagnosis of either DVT, PE or both).
* Any patient receiving crizanlizumab therapy for SCD or that has received crizanlizumab within the past 30 days of D0 of study.
* Have a significant medical condition that confers an unacceptable risk to participating in the study, and/or that could confound the interpretation of the study data. Such significant medical conditions include, but are not limited to the following:

  1. History of recent (within 3 months prior to signing informed consent) congestive heart failure; myocardial infarction or unstable angina pectoris; hemorrhagic, embolic, or thrombotic stroke.
  2. Active infection requiring the use of parenteral antimicrobial agents or Grade greater than or equal to 3 in severity (per National Cancer Institute Common Terminology Criteria for Adverse Events v5.0) within 2 months prior to the first dose of study drug.
  3. Active viral infection as evidenced by testing positive for hepatitis B surface antigen or hepatitis C virus (HCV) antibody (Ab) with signs of active hepatitis B or C virus infection. If the subject is positive for HCV Ab, a reverse transcriptase-polymerase chain reaction test will be conducted. Subjects with hepatitis C may be rescreened after receiving appropriate hepatitis C treatment.
  4. Testing positive for human immunodeficiency virus (HIV) 1 or 2 Ab with evidence for ongoing active infection (i.e., CD4 count <400/microL and viral load >100,000 copies/mL) on antiretroviral therapy.
  5. Active acute inflammatory disorders rheumatoid arthritis or systemic lupus erythematosus on disease modifying therapy.
  6. Diabetes mellitus judged to be under poor control by the Investigator evidenced by a single fasting sugar value >250 gm/dl or requiring >3 antidiabetic agents, including insulin (all insulins are considered 1 agent); use of insulin per se is not exclusionary.
  7. History of any primary malignancy, with the exception of curatively treated nonmelanomatous skin cancer; curatively treated cervical or breast carcinoma in situ; or other primary tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years.
  8. Any injury or medical condition that, in the judgement of the Investigator would prevent the subject from participating in the study.
* Have a prior bone marrow or stem cell transplant.

INCLUSION OF VULNNERABLE PARTICIPANTS:

Vulnerable subjects will not be included in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun S Shet, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Lizarralde-Iragorri MA, Parachalil Gopalan B, Merriweather B, Brooks J, Hill M, Lovins D, Pierre-Charles R, Cullinane A, Dulau-Florea A, Lee DY, Villasmil R, Jeffries N, Shet AS. Isoquercetin for thromboinflammation in sickle cell disease: a randomized double-blind placebo-controlled trial. Blood Adv. 2024 Jan 9;8(1):172-182. doi: 10.1182/bloodadvances.2023011542. PMID 38157227
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-H-0137.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Sickle Cell Disease Receiving Isoquercetin: Isoquercetin given 1000 mg, once daily by mouth for 28 days in participants with Sickle Cell Disease.
- Participants With Sickle Cell Disease Receiving Placebo: Placebo given once daily, by mouth for 28 days in participants with Sickle Cell Disease.
Period: Overall Study
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Started | 23 | 23
Completed | 22 | 22
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Randomized but did not receive Isoquercetin | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 22 | 20 | 42
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 22 | 43
  White | 0 | 0 | 0
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Plasma Soluble P-selectin Level
Description: Mean change in plasma soluble P-selectin level comparing the baseline versus IQ or placebo.
Time Frame: Baseline and Day 28
Population: One patient in the isoquercetin arm was randomized but withdrawn from the study before any treatment and did not provide baseline soluble P-selectin measurement nor contribute to this analysis. One patient in the placebo arm provided baseline soluble P-selectin and their change in P-selectin was obtained via a multiple imputation procedure. 45 participants (22 isoquercetin and 23 placebo) contributed to the analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 22 | 23
ng/ml | 0.74 (6.53) | 0.10 (4.54)
Statistical Analysis 1: Comparison: Participants With Sickle Cell Disease Receiving Isoquercetin vs Participants With Sickle Cell Disease Receiving Placebo; Test type: Superiority; p = 0.64, ANCOVA with Multiple Imputation

2. Secondary Outcome: Mean Change in Plasma Protein Disulfide Isomerase Activity
Description: Mean Change in Plasma Protein Disulfide Isomerase Activity comparing baseline and end of study
Time Frame: Baseline and 28 days
Population: Analysis includes only participants that completed study
Measure: Mean (Standard Deviation); unit: pMoles/min/µL
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 22 | 22
pMoles/min/µL | -3.13 (10.91) | 1.95 (9.34)

3. Secondary Outcome: Median Change of Tissue Factor Vesicle Number
Description: Median change of Tissue Factor Vesicle Number comparing baseline and end of study
Time Frame: Baseline and Day 28
Population: Analysis includes only participants that completed study
Measure: Median (Inter-Quartile Range); unit: microvesicles/mL
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 22 | 22
microvesicles/mL | 39 [-115 to 1296] | -382 [-1090 to 86]

4. Secondary Outcome: Mean Change in Tissue Factor Vesicle Procoagulant Activity
Description: Mean change in tissue factor vesicle procoagulant activity comparing baseline and end of study
Time Frame: Baseline and Day 28
Population: Analysis includes only participants that completed study
Measure: Mean (Standard Deviation); unit: Picomoles
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 22 | 22
Picomoles | -427 (1868) | -43 (1404)

5. Secondary Outcome: Mean Change in D-Dimer
Description: Mean Change in D-Dimer comparing baseline and end of study
Time Frame: Baseline and Day 28
Population: Analysis includes only participants that completed study
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 22 | 22
mcg/mL | 0.15 (0.92) | 0.28 (1.18)

6. Secondary Outcome: Mean Change in Vascular Cell Adhesion Molecule
Description: Mean Change in Vascular Cell Adhesion Molecule (inflammation marker) comparing baseline to Day 28
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 22 | 22
ng/mL | -22.43 (291.42) | -38.15 (180.24)

7. Secondary Outcome: Median Relative Blood Flow Index (rBFI) Determined by Near-infrared Spectroscopy (NIRS)
Description: Median Relative Blood Flow Index (rBFI) determined by Near-infrared spectroscopy (NIRS).
  Near-infrared spectroscopy (NIRS) is a noninvasive technology that measures blood flow by directing near-infrared light into tissue, collects scattered light due to red blood cell movements using photodiodes, and calculates the blood flow index (BFI) using the correlation diffusion equation (CDE). Briefly, participants were seated upright and NIRS probe and a blood pressure cuff was placed on the right arm and resting baseline data was collected for three minutes followed by occlusion of the blood flow for three minutes and reperfusion recorded for three minutes. The post-occlusion hyperemic reperfusion response represented as the relative Blood Flow Index (rBFI) is determined by normalizing the maximal change in light absorption following occlusion (dBFI) by the corresponding time interval (dt); (rBFI = dBFI/dt; unit (cm^2/s)/s)].
Time Frame: Day 28
Population: Analysis includes those participants that completed the end of study Near-infrared spectroscopy (NIRS) procedure.
Measure: Median (Inter-Quartile Range); unit: (cm2/s)/s
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 5 | 7
(cm2/s)/s | 0.00000000082 [0.00000000046 to 0.0000000021] | 0.00000000037 [0.00000000021 to 0.0000000013]
Statistical Analysis 1: Comparison: Participants With Sickle Cell Disease Receiving Isoquercetin vs Participants With Sickle Cell Disease Receiving Placebo; Test type: Superiority; p = 0.149, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Mean Percent Adherence to Study Drug
Description: Mean percent adherence to study drug. Adherence was defined as number of study drug pills participant took divided by number of study drug pills dispensed multiplied by 100.
Time Frame: Baseline and Day 28
Population: Analysis includes only participants that completed study
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 22 | 22
percentage of adherence | 96.2 (13.9) | 97.2 (4.7)

9. Secondary Outcome: Number of Adverse Events Grade 2 and Above
Description: Number of adverse events Grade 2 and above using Common Terminology Criteria for Adverse Events (CTCAE) 5.0
Time Frame: Up to Day 56
Measure: Number; unit: Adverse Events
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 23 | 23
Adverse Events
  Grade 2 | 8 | 9
  Grade 3 and 4 | 1 | 2
  Serious Adverse Events | 8 | 6

10. Secondary Outcome: Number of Participants That Tolerated Study Drug
Description: Number of participants that tolerated study drug for full duration of study
Time Frame: Up to day 28
Population: Analysis includes only participants that completed study
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
Number analyzed (Participants) | 22 | 22
Participants | 22 | 22

ADVERSE EVENTS:
Time Frame: Up to 56 days
Description: Investigators will assess the occurrence of adverse events (AEs) and serious adverse events (SAEs) at all patient evaluation time points during the study. Grade 2 and above plus clinically significant laboratory abnormalities whether volunteered by the patient, discovered by study personnel during questioning, or detected through physical examination, clinically significant laboratory test, or other means will be recorded.
Arm/Group | Participants With Sickle Cell Disease Receiving Isoquercetin | Participants With Sickle Cell Disease Receiving Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 6/23 | 4/23
Other Adverse Events (participants affected / at risk) | 9/23 | 11/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Sickle Cell Disease Receiving Isoquercetin (N=23) | Participants With Sickle Cell Disease Receiving Placebo (N=23)
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 5 (5) | 4 (5)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Sickle Cell Disease Receiving Isoquercetin (N=23) | Participants With Sickle Cell Disease Receiving Placebo (N=23)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic sickle cell pain (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Headache (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT04514510/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT04514510/SAP_003.pdf
  • Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT04514510/ICF_001.pdf